CLINICAL TRIAL: NCT03707886
Title: Pain SMART: Shared Medical Appointments to Refocus Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Collaborators: VISN1 Career Development Award Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 02103-0001
Record Dates: First submitted 2018-08-28; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Chronic Pain
Keywords: chronic pain; shared medical appointment; veterans
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain SMART (Intervention Arm) (Experimental): The Intervention Arm will be invited to participate in a one-time group intervention, Pain SMART
  Interventions: Behavioral: Pain SMART
- Minimally Enhanced Usual Care (Placebo Comparator): The Minimally Enhanced Usual Care group will receive educational information via mail.
  Interventions: Other: minimally enhanced usual care

INTERVENTIONS:
Behavioral: Pain SMART — Pain SMART is a brief, one-visit shared medical appointment where providers in primary care and a behavioral health specialist (e.g., a psychologist) meet with a group of patients with chronic pain to discuss pain management approaches.
  Arms: Pain SMART (Intervention Arm)
Other: minimally enhanced usual care — The minimally enhanced usual care group will receive educational information via mail about non-pharmacological approaches to pain management.
  Arms: Minimally Enhanced Usual Care

SUMMARY:
The proposed study will test whether a shared medical appointment for Veterans with chronic pain is feasible and acceptable to veteran patients and their providers. The shared medical appointment, called Pain SMART (Shared Medical Appointments to Refocus Treatment), is a brief, one-visit shared medical appointment where providers in primary care and a behavioral health specialist (e.g., a psychologist) meet with a group of patients with chronic pain. The overall goal of Pain SMART is to improve pain care for Veterans. Veterans will be randomized in equal numbers to either attend a Pain SMART visit or to receive educational information in the mail. The primary outcome of this pilot study is whether or not the shared medical appointment is feasible and acceptable to patients and providers.

DETAILED DESCRIPTION:
Objectives: The primary purpose of this study is to understand the feasibility and acceptability of a shared medical appointment for patients with chronic pain called Pain SMART (Shared Medical Appointments to Refocus Treatment).

Intervention: The overall goal of Pain SMART is to increase the use of evidenced-based pain management strategies including pain self-management and other non-pharmacological pain management approaches. Pain SMART is a brief one-visit shared medical appointment delivered by primary care team members (e.g., primary care providers) and a behavioral health specialist (e.g., a clinical health psychologist). Pain SMART uses motivational interviewing to enhance effective and mutually rewarding communication among providers and Veterans to increase pain self-management, including uptake of non-pharmacological approaches to pain management, to ultimately enhance quality of care and Veteran functioning.

Study Participants: Primary care providers/staff will be recruited to participate in Pain SMART visits as shared medical appointment facilitators. Additionally, up to 80 veterans with chronic pain will be recruited.

Research Design: This study is a randomized pilot study in which Veteran participants are randomized to attend Pain SMART or to a minimally enhanced usual care condition (i.e., receive an educational brochure via mail). Veteran participants will be randomized in equal numbers to both conditions. Data collected from Veteran participants at baseline and three months following baseline; data will also be collected from primary care participants regarding their experience with Pain SMART. Data collection will include quantitative measures (e.g., information regarding pain and pain management approaches used) and qualitative measures (e.g., interviews about participants' experiences with Pain SMART).

ELIGIBILITY:
Veteran Inclusion Criteria:

* Receives primary care from provider at VA Connecticut who is participating in the study
* Prescribed an opioid for chronic pain

Veteran Exclusion Criteria:

* Active suicidal ideation
* Psychotic disorder
* Active consult to opioid reassessment clinic at VA Connecticut

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of participant recruitment | 3 months
  ability to recruit Veterans to enroll in the study and attend group, as evidenced by randomizing 80 veterans over the study period and by having at least 60% of veterans randomized to attend the group show up to to the group

SECONDARY OUTCOMES:
Pain management strategies used - Chronic Pain Coping Inventory | 3 months
  The chronic pain coping inventory measures the use of pain self-management strategies (e.g., activity pacing)

OTHER OUTCOMES:
Pain management strategies used - Self-reported use of pain management strategies | 3 months
  We have developed a measure that asks participants if they have tried any pain management strategies in the past three months (e.g., acupuncture, cognitive behavioral therapy).

CONTACTS AND LOCATIONS:
Locations (1):
- Va Connecticut Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No